CLINICAL TRIAL: NCT02742428
Title: Preoperative Slow Ascites Drainage Versus Standard Care for Patients With Proven or Suspected Advanced Ovarian Cancer - a Hemodynamic Impact on Systemic Circulation, Patient's Nutritional Status and Quality of Life: a Randomized Trial.
Brief Title: Preoperative Ascites Drainage Versus Standard Care for Patients With Advanced Ovarian Cancer
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol will be discussed and consulted. Potentially will resume.
Sponsor: Gdynia Oncology Center (Other Government)
Responsible Party: Principal Investigator, Maciej Stukan, MD, PhD, Dr, Gdynia Oncology Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO-2
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Ascites; Ovarian Epithelial Cancer; Malnutrition
MeSH Terms: conditions — Ascites; Carcinoma, Ovarian Epithelial; Malnutrition | interventions — Interviews as Topic; Quality of Life; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascites drainage before surgery. (Experimental): A group of patients with (or suspected for) advanced ovarian cancer and significant ascites. An indwelling catheter insertion into abdominal cavity and slow, systematic ascites evacuation for 7 or more days before surgery (if it cannot be scheduled immediately) will be performed. Patients will undergo an interview, will be asked to fill in questionnaires concerning a quality of life and nutritional status. If available noninvasive bioimpedance analysis will be performed and 2ml of blood will be taken for serum prealbumin concentration evaluation. If possible 20ml of ascitic fluid will be taken for cytology examination.
  Interventions: Device: Systematic ascites evacuation; Behavioral: Interview.; Behavioral: Quality of life.; Behavioral: Nutritional status.
- Observation. (Other): A group of patients with (or suspected for) advanced ovarian cancer and significant ascites. A standard of care: observation or acute paracentesis (>5000ml) will be performed while waiting for the surgery (if it cannot be scheduled immediately). Patients will undergo an interview, will be asked to fill in questionnaires concerning a quality of life and nutritional status. If available noninvasive bioimpedance analysis will be performed and 2ml of blood will be taken for serum prealbumin concentration evaluation. If possible 20ml of ascitic fluid will be taken for cytology examination.
  Interventions: Procedure: Acute paracentesis.; Behavioral: Interview.; Behavioral: Quality of life.; Behavioral: Nutritional status.

INTERVENTIONS:
Device: Systematic ascites evacuation — Systematic ascites evacuation via indwelling catheter inserted into abdominal cavity, sutured to the skin. Drainage performed by the patient, on demand with day limit of 2000ml, in ambulatory settings.
  Arms: Ascites drainage before surgery.
Procedure: Acute paracentesis. — Evacuation of a large (>5000ml) volume of ascites via single abdominocentesis. Allowed in observational arm only, in case of acute symptoms concerned with ascites.
  Arms: Observation.
Behavioral: Interview. — Interview according to provided chart in order to collect data concerning symptoms, co-morbidities.
Behavioral: Quality of life. — Patients will be asked to fill in a quality of life questionnaire (EORTC-C15-PAL) before randomization and 7 days later.
Behavioral: Nutritional status. — Patients will be asked to fill in (together with a physician) a questionnaire to assess risk of malnutrition (SGA) before randomization and 7 days later.

SUMMARY:
Patients with significant ascites and advanced ovarian cancer (AOC), undergoing complex, cytoreductive surgery are at risk of malnutrition, poor quality of life and the risk of hypo- or hypervolemia in a perioperative period. All these factors may cause hemodynamic consequences during anesthesia and surgery, and elevate the risk of morbidity and mortality.

The objective of the study is to evaluate, whether slow ascites evacuation for a few days before the surgery for AOC, could 1) influence the hemodynamic consequences of ascites on systemic circulation in patients undergoing surgery, 2) improve patient's quality of life and 3) ability to feed correctly before treatment starts, and thus lower the risk of perioperative morbidity.

Eligible patients are those with significant ascites, diagnosed or suspected for AOC, who are scheduled for primary surgery (both upfront cytoreduction or laparoscopic evaluation before neoadjuvant chemotherapy), that cannot be performed within next 7 or more days, for any reason. Patients will be asked to fill in quality of life questionnaire (QLQ). Clinical data, a Subjective Global Assessment (SGA) will be recorded. Patients will be randomized to either intervention arm A - insertion of vascular catheter into abdominal cavity and slow, systematic, daily ascites evacuation, or to observation arm B - standard of care with just observation (acute large volume (>5000ml) paracentesis allowed if needed). Patients in both groups will be encouraged to use oral nutritional support. Randomization will be open, 1:1, for every eligible, consecutive patient. After 7 days patients will be interviewed, asked to fill in QLQ, patient's experience on the treatment survey, a SGA will be recorded. During the first hour of the surgery hemodynamic data from anethetic charts will be recorded along with other clinical data concerning patient's characteristics, surgery details and 30-day postoperative follow-up. A template is provided.

The hypothesis of the study is that slow, systematic ascites evacuation few days before surgery for advanced ovarian cancer can facilitate hemodynamic control of systemic circulation of patients undergoing surgery, and improve patients' quality of life, feeding ability before treatment starts. Secondary we would expect lower risk of perioperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* patients with significant ascites and suspected ovarian cancer scheduled for upfront cytoreductive surgery, or diagnostic laparoscopy and neoadjuvant chemotherapy, and the surgery is planned to be performed in at least 7 days,
* signed informed consent of the patient.

Exclusion Criteria:

* ascites not of malignant origin,
* low volume ascites,
* other then primary ovarian malignancy suspected,
* suspected or clinically apparent infection especially at the site of planned drainage placement,
* no patient's consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Changes in median arterial pressure (MAP) during anesthesia. | 1 hour
  Changes (minimal and maximal) in median arterial pressure during 1st hour of anesthesia during cytoreductive surgery for advanced ovarian cancer - comparison of two groups: with and without preoperative ascites drainage. MAP calculation - MAP = [(2 x diastolic)+systolic] / 3.
Volume of intravenous fluids transfused. | 1 hour
  Volume of intravenous fluids transfused during the 1st hour of cytoreductive surgery for advanced ovarian cancer - comparison of two groups: with and without preoperative ascites drainage.
Number of participants who required vasoconstrictors. | 1 hour
  Need for using vasoconstrictors during 1st hour of cytoreductive surgery for advanced ovarian cancer - comparison of two groups: with and without preoperative ascites drainage.
Changes in Heart Rate (HR). | 1 hour
  Changes in HR (minimal and maximal) during 1st hour of anesthesia during cytoreductive surgery for advanced ovarian cancer - comparison of two groups: with and without preoperative ascites drainage.

SECONDARY OUTCOMES:
Changes in feeding ability. | 7 days
  Evaluation of changes in feeding ability before the treatment starts, according to Subjective Global Assesment survey - comparison of two groups: with and without preoperative ascites drainage.
Changes in patients' quality of life. | 7 days
  To note any changes in quality of life evaluated with standardized quality of life questionnaire.

OTHER OUTCOMES:
Number of adverse events concerned with indwelling catheter insertion. | 7 days
  Number of adverse events concerned with catheter insertion for ascites drainage.
Number of participants correctly diagnosed with ovarian cancer based on ascitic fluid cytology. | 1 day
  Ascitis fluid collected for cytology examination. The accuracy of ascitic fluid cytology in diagnosing ovarian cancer.
Changes in Extracellular Fluid (ECF) and Intracellular Fluid (ICF). | 7 days
  Changes in body fluid balance measured with bioimpedance analysis tools and defined with ECF and ICF. Parameters will be recorded at randomization, before surgery, and during the 1st hour of the anesthesia.
Changes in Phase Angle (PA). | 7 days
  Changes in nutritional status measured with bioimpedance analysis tools and defined with PA. Parameters will be recorded at randomisation and before the surgery.
Changes in prealbumin concentration. | 7 days
  Changes in nutritional status measured with prealbumin plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Stukan, MD, PhD, Principal Investigator — Gdynia Oncology Center
Locations (1):
- Gdynia Oncology Center, Gdynia, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunsicker O, Fotopoulou C, Pietzner K, Koch M, Krannich A, Sehouli J, Spies C, Feldheiser A. Hemodynamic Consequences of Malignant Ascites in Epithelial Ovarian Cancer Surgery*: A Prospective Substudy of a Randomized Controlled Trial. Medicine (Baltimore). 2015 Dec;94(49):e2108. doi: 10.1097/MD.0000000000002108. PMID 26656336
- [Background] Feldheiser A, Braicu EI, Bonomo T, Walther A, Kaufner L, Pietzner K, Spies C, Sehouli J, Fotopoulou C. Impact of ascites on the perioperative course of patients with advanced ovarian cancer undergoing extensive cytoreduction: results of a study on 119 patients. Int J Gynecol Cancer. 2014 Mar;24(3):478-87. doi: 10.1097/IGC.0000000000000069. PMID 24463641
- [Result] Stukan M, Lesniewski-Kmak K, Wroblewska M, Dudziak M. Management of symptomatic ascites and post-operative lymphocysts with an easy-to-use, patient-controlled, vascular catheter. Gynecol Oncol. 2015 Mar;136(3):466-71. doi: 10.1016/j.ygyno.2014.11.073. Epub 2014 Nov 28. PMID 25434633
- [Result] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for pre- and intra-operative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part I. Gynecol Oncol. 2016 Feb;140(2):313-22. doi: 10.1016/j.ygyno.2015.11.015. Epub 2015 Nov 18. No abstract available. PMID 26603969